CLINICAL TRIAL: NCT03075566
Title: Clinical and Biochemical Markers in Coronary Artery Disease
Brief Title: Coronary Artery Disease: a Case- Control Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nadia Bouzidi, PhD (Other)
Responsible Party: Sponsor-Investigator, Nadia Bouzidi, PhD, Bouzidi Nadia, PhD, University of Monastir
Organization: University of Monastir (Other)
Other Study IDs: 1500170
Record Dates: First submitted 2017-02-05; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; risk factors; inflammation; biomarkers; atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Inflammation; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: Healthy subjects — - 207 healthy subjects were donors,(33.2±12.2 years) recruited from the Blood Bank Department of the University Hospital (Mahdia, Tunisia).
Biological: Patients — - 310 subjects with CAD (60.3±11.0 years) were admitted to the Department of Cardiology, University Hospital (Monastir, Tunisia).

SUMMARY:
Atherosclerosis is a chronic inflammatory condition, which is associated by the involvement of several pathological events, and alteration in the serum levels of pro- and anti-inflammatory, and lipid markers.

The investigators evaluated the contribution of serum biomarkers levels to the pathogenesis of coronary artery disease, namely their association with risk factors, clinical presentation, extent and severity of atherosclerotic changes accompanying coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Disease

Exclusion Criteria:

* Severe respiratory disease
* Liver disease
* kidney disease
* Inflammatory diseases (infections, autoimmune disorders, malignancy).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 310 patients with Coronary Artery Disease
  * 207 healthy subjects
Sampling Method: Probability Sample
Enrollment: 517 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical parameters | 1 Days
  * Glucose (mmol/l), urae (mmol/l), creatinin (µmol/l), total cholesterol (mmol/l), high density lipoprotein cholesterol, HDL-C (mmol/l), triglycerides (mmol/l), lipoprotein(a) (g/l), apolipoproteins, apo (g/l) were measured only once in each patient at admission, before angiography and in each control group participant using the COBAS INTEGRA 400 chemical analyzer (Roche Diagnostic, Germany).
  * Troponin I (ng/ml), creatine kinase (CK) (UI/L), creatine kinase MB Isoenzyme (CK-MB)(UI/L), glutamic-oxaloacetic transaminase (ASAT) (UI/L) were measured using the COBAS INTEGRA 400 chemical analyzer (Roche Diagnostic, Germany). Only one measure was performed for each participant regarding all these parameters.
  * Light density lipoprotein cholesterol, LDL-C (mmol/l) was estimated using the Friedewald equation. Only one measure was performed for each participant.
  * Values which were out of the confidence range were considered as abnormal values.
Inflammatory markers | 2 Days
  * Serum Amyloid A (SAA) (mg/l) was measured using the BN Prospec, Siemens.
  * High sensitivity C reactive protein, hsCRP (mg/l) was measured using the COBAS INTEGRA 400 chemical analyzer (Roche Diagnostic, Germany).
  * Activin A (pg/ml) was quantified at 450nm using a commercially available ELISA kit (AbFrontier, Young In Frontier Co., Ltd, Korea). Only one measure was performed for each participant.
  * Interleukin-6 (pg/ml) was measured using a Cobas E601 analyzer (Roche Diagnostics, Germany). Only one measure was performed for each participant.
  * Values which were out of the confidence range were considered as abnormal values.

CONTACTS AND LOCATIONS:
Overall Officials: Salima Ferchichi, Pr, Study Director — University of Monastir, Faculty of Pharmacy of Monastir, Tunisia
Locations (1):
- Faculty of Pharmacy, Monastir, Ibn Sina Street, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouzidi N, Gamra H. Relationship between serum interleukin-6 levels and severity of coronary artery disease undergoing percutaneous coronary intervention. BMC Cardiovasc Disord. 2023 Nov 28;23(1):586. doi: 10.1186/s12872-023-03570-8. PMID 38017432